CLINICAL TRIAL: NCT00509288
Title: Phase II Study of Metastatic Melanoma Using Lymphodepleting Conditioning Followed by Infusion of Anti-MART-1 F5 TCR-Gene Engineered Lymphocytes
Brief Title: Phase II Study of Metastatic Melanoma With Lymphodepleting Conditioning and Infusion of Anti-MART-1 F5 TCR-Gene-Engineered Lymphocytes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070175; 07-C-0175
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Melanoma; Skin Cancer
Keywords: Refractory; Gene Therapy; HLA-A2 Positive; Stage IV Melanoma; Melanoma; Skin Cancer; Malignant Melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anti-MART-1 F5 TCR PBL + HD IL-2 (Experimental): Patients treated with peripheral blood lymphocytes (PBL)
  Interventions: Biological: autologous anti-MART-1 F5 T-cell receptor; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Aldesleukin
- anti-MART-1 F5 TCR TIL + HD IL-2 (Experimental): Patients treated with TIL (tumor infiltrating lymphocytes).
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Aldesleukin; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered tumor infiltrating lymphocytes

INTERVENTIONS:
Biological: autologous anti-MART-1 F5 T-cell receptor — Autologous anti-MART-1 F5 T-cell receptor gene-engineered tumor infiltrating lymphocytes.
  A minimum of approximately 5 X 10^8 cells will be given up to 3x10^11 anti-MART-1 F5 TCR engineered TIL or PBL.
  Arms: anti-MART-1 F5 TCR PBL + HD IL-2
Drug: Cyclophosphamide — Day -7 to -5: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Other Names: Cytoxan
Drug: Fludarabine — Day -5 to 1: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days
  Other Names: Fludara
Biological: Aldesleukin — Day 0: Cells will be infused intravenously (i.v.). Patients will receive up to 3x10e^11 (with a minimum of 5x10e^8 cells) anti-MART-1 F5 TCR engineered TIL or PBL Aldesleukin (based on total body weight) 720,000 IU/kg intravenous (IV) over 15 minute every eight hours beginning within 24 hours of cell infusion
  Other Names: IL-2
Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered tumor infiltrating lymphocytes
  Arms: anti-MART-1 F5 TCR TIL + HD IL-2

SUMMARY:
Background:

* Human peripheral blood lymphocytes have been engineered to express a T-cell receptor (TCR) that recognizes a blood type,HLA-A 0201 (human leukocyte antigen) derived from the gp100 protein. A retroviral vector was constructed that can deliver the T-cell receptor (TCR) to cells.
* Patients' cells will be converted into cells able to recognize and fight melanoma tumors.

Objectives:

* To determine whether TCR-engineered lymphocytes can be put in cells removed from patients' tumors or blood and then reinfused, with the purpose of shrinking tumors.
* To evaluate safety and effectiveness of the treatment.

Eligibility:

* Patients 18 years of age or older with metastatic cancer melanoma (cancer that has spread beyond the original site).
* Patient's leukocyte antigen type is HLA-A 0201.

Design:

-Patients undergo the following procedures:

* Leukapheresis (on two occasions). This is a method of collecting large numbers of white blood cells. The cells obtained in the first leukapheresis procedure are grown in the laboratory, and the anti-MART-1 protein is inserted into the cells using an inactivated (harmless) virus in a process called retroviral transduction. Cells collected in the second leukapheresis procedure are used to evaluate the effectiveness of the study treatment.
* Chemotherapy. Patients are given chemotherapy through a vein (intravenously, IV) over 1 hour for 2 days to suppress the immune system so that the patient's immune cells do not interfere with the treatment.
* Treatment with anti-melanoma antigen recognized by T-cells (MART)-1. Patients receive an intravenous (IV) infusion of the treated cells containing anti-MART-1 protein, followed by infusions of a drug called IL-2 (aldesleukin), which helps boost the effectiveness of the treated white cells.
* Patients are given support medications to prevent complications such as infections.
* Patients may undergo a tumor biopsy (removal of a small piece of tumor tissue).
* Patients are evaluated with laboratory tests and imaging tests, such as CT (computed tomography) scans, 4 to 6 weeks after treatment and then once a month for 3 to 4 months to determine the response to treatment.
* Patients have blood tests at 3, 6, and 12 months and then annually for 5 years.

DETAILED DESCRIPTION:
Background:

* We have engineered human TIL (tumor infiltrating lymphocytes) and peripheral blood lymphocytes (PBLs) to express an anti-MART-1 T-cell receptor that recognizes an HLA-A*0201 restricted epitope derived from the TIL clone DMF5.
* We constructed a single retroviral vector that contains both alpha and beta chains and can mediate genetic transfer of this TCR with high efficiency without the need to perform any selection.
* In co-cultures with HLA-A*0201 positive melanoma, anti-MART-1 F5 TCR transduced T cells secreted significant amount of interferon (IFN)-gamma (but no significant secretion was observed in control co-cultures with cell lines.
* The anti-MART-1 F5 TCR transduced T-cells could efficiently kill HLA-A*0201 positive tumors. There was little or no recognition of normal fibroblasts cells.
* This TCR is over 10 times more reactive with melanoma cells than the MART-1 TCR that mediated tumor regression in two patients with metastatic melanoma.

Objectives:

Primary objectives:

-Determine if the administration of anti-MART-1 F5 TCR -engineered peripheral blood lymphocytes (PBL) or tumor infiltrating lymphocytes (TIL) and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic melanoma.

Secondary objectives:

* Determine the in vivo survival of TCR gene-engineered cells.
* Determine the toxicity profile of this treatment regimen.

Eligibility:

Patients who are HLA-A 0201 positive and 18 years of age or older must have:

* metastatic melanoma;
* previously received and have been a non-responder to or recurred after aldesleukin;
* normal values for basic laboratory values.

Patients may not have:

* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* severe hypersensitivity to any of the agents used in this study;
* contraindications for high dose aldesleukin administration.

Design:

* If TIL can be obtained and grown, but are non-reactive, patients will be assigned to receive TIL transduced with the anti-MART-1 F5 TCR retroviral vector. If TIL cannot be obtained, PBMC will be obtained by leukapheresis (approximately 5 X 10(9) cells) and cultured in the presence of anti-CD3 (OKT3) and aldesleukin and transduced with the anti-MART-1 F5 TCR retroviral vector. If TIL cells are reactive to autologous tumor or major histocompatibility complex (MHC)-matched tumor cells or PBL cannot be grown, patients will not be treated on this protocol.
* Transduction is initiated by exposure of approximately 10(8) to 5 times 10(8) cells to retroviral vector supernatant containing the anti-MART-1 F5 TCR genes. These transduced cells will be expanded and tested for their anti-tumor activity.
* Once engineered lymphocytes are demonstrated to be biologically active according to the strict criteria outlined in the Certificate of Analysis, patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene transduced cells plus IV aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses).
* Patients will undergo complete evaluation of tumor with physical examination, CT of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.
* The study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled into each of two cohorts. If 0 or 1 of the 21 patients per cohort experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled in that cohort have a clinical response, then accrual to that cohort will continue until a total of 41 evaluable patients have been enrolled in that cohort.
* The objective will be to determine in two cohorts if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-MART-1 F5 TCR-gene engineered lymphocytes (TIL and PBL) is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% PR (partial response) + CR (complete response) rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic melanoma with measurable disease
  2. Previously received high dose IL-2 (aldesleukin) and have been either non-responders (progressive disease) or have recurred.
  3. Positive for MART-1 by immunohistochemistry (IHC)
  4. Greater than or equal to 18 years of age.
  5. Willing to sign a durable power of attorney
  6. Able to understand and sign the Informed Consent Document
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  8. Life expectancy of greater than three months.
  9. Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
  10. Patients must be human leukocyte antigen (HLA-A)*0201 positive
  11. Serology:

  <!-- -->

  1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
  3. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

  l. Hematology:
  1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
  2. White blood cell (WBC) (greater than 3000/mm^3).
  3. Platelet count greater than 100,000/ mm^3.
  4. Hemoglobin greater than 8.0 g/dl.

  m. Chemistry:
  1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
  2. Serum creatinine less than or equal to 1.6 mg/dl.
  3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

  n. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

  o. Six weeks must have elapsed since prior anti-CTLA4 antibody therapy to allow antibody levels to decline.

  p. Patients who have previously received anti-CTLA4 antibody must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Patients with reactive TIL (IFN-gamma release greater than 200 pg/mL) available based on overnight co-culture assay with autologous tumor or MHC-matched tumor cells.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
6. Systemic steroid therapy.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms.
9. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45 percent.
10. Documented LVEF of less than or equal to 45 percent tested in patients with:

    * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block.
    * Age greater than or equal to 60 years old.
11. Documented forced expiratory volume 1 (FEV1) less than or equal to 60 percent predicted tested in patients with:

    * A prolonged history of cigarette smoking (20 pk/yrs of smoking).
    * Symptoms of respiratory dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Sakaguchi K, Appella E, Yannelli JR, Adema GJ, Miki T, Rosenberg SA. Identification of a human melanoma antigen recognized by tumor-infiltrating lymphocytes associated with in vivo tumor rejection. Proc Natl Acad Sci U S A. 1994 Jul 5;91(14):6458-62. doi: 10.1073/pnas.91.14.6458. PMID 8022805
- [Derived] Abate-Daga D, Hanada K, Davis JL, Yang JC, Rosenberg SA, Morgan RA. Expression profiling of TCR-engineered T cells demonstrates overexpression of multiple inhibitory receptors in persisting lymphocytes. Blood. 2013 Aug 22;122(8):1399-410. doi: 10.1182/blood-2013-04-495531. Epub 2013 Jul 16. PMID 23861247
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0175.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-MART-1 F5 TCR PBL + HD IL-2: Patients treated with peripheral blood lymphocytes (PBL). A minimum of approximately 5 X 10^8 cells will be given up to 3x10^11 anti-MART-1 F5 TCR engineered TIL or PBL. Day -7 to -5: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr. Day -5 to 1: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days. Day 0: Cells will be infused intravenously (i.v.). Patients will receive up to 3x10e^11 (with a minimum of 5x10e^8 cells) anti-MART-1 F5 TCR engineered TIL or PBL Aldesleukin (based on total body weight) 720,000 IU/kg intravenous (IV) over 15 minute every eight hours beginning within 24 hours of cell infusion.
- Anti-MART-1 F5 TCR TIL + HD IL-2: Patients treated with tumor infiltrating lymphocytes (TIL). A minimum of approximately 5 X 10^8 cells will be given up to 3x10^11 anti-MART-1 F5 TCR engineered TIL or PBL. Day -7 to -5: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr. Day -5 to 1: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days Day 0: Cells will be infused intravenously (i.v.). Patients will receive up to 3x10e^11 (with a minimum of 5x10e^8 cells) anti-MART-1 F5 TCR engineered TIL or PBL Aldesleukin (based on total body weight) 720,000 IU/kg intravenous (IV) over 15 minute every eight hours beginning within 24 hours of cell infusion.
Period: Overall Study
Arm/Group | Anti-MART-1 F5 TCR PBL + HD IL-2 | Anti-MART-1 F5 TCR TIL + HD IL-2
Started | 21 | 3
Completed | 21 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Anti-MART-1 F5 TCR TIL + HD IL-2: Patients treated with tumor infiltrating lymphocytes (TIL).
- Total: Total of all reporting groups
Arm/Group | Anti-MART-1 F5 TCR PBL + HD IL-2 | Anti-MART-1 F5 TCR TIL + HD IL-2 | Total
Number analyzed (Participants) | 21 | 3 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 3 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.0) | 48.0 (21.7) | 46.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 12 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 3 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 3 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tumor Regression.
Description: Tumor regression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 7/5/07-4/23/09
Measure: Number; unit: Participants
Arm/Group | Anti-MART-1 F5 TCR PBL + HD IL-2 | Anti-MART-1 F5 TCR TIL + HD IL-2
Number analyzed (Participants) | 21 | 3
Participants
  Complete Response | 0 | 0
  Partial Response | 6 | 0
  Progressive Disease | 15 | 2
  Stable Disease | 0 | 0

2. Secondary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed listing of adverse events, see the adverse event module.
Time Frame: 57 months
Measure: Number; unit: Participants
Arm/Group | Anti-MART-1 F5 TCR PBL + HD IL-2 | Anti-MART-1 F5 TCR TIL + HD IL-2
Number analyzed (Participants) | 21 | 3
Participants | 21 | 3

ADVERSE EVENTS:
Arm/Group | Anti-MART-1 F5 TCR PBL + HD IL-2 | Anti-MART-1 F5 TCR TIL + HD IL-2
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/3
Other Adverse Events (participants affected / at risk) | 21/21 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-MART-1 F5 TCR PBL + HD IL-2 (N=21) | Anti-MART-1 F5 TCR TIL + HD IL-2 (N=3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-MART-1 F5 TCR PBL + HD IL-2 (N=21) | Anti-MART-1 F5 TCR TIL + HD IL-2 (N=3)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Hearing: patients with/without baseline audiogram (Ear and labyrinth disorders) | 10 (11) | 0 (0)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (5) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 11 (12) | 3 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 20 (22) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 20 (25) | 3 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 20 (23) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 20 (22) | 3 (3)
Prolonged QTc interval (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 11 (12) | 0 (0)
Vasovagal episode (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 3 (3) | 0 (0)
Hypotension (Cardiac disorders) | 10 (14) | 2 (2)
left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Constitutional Symptoms-Other (Specify, insomnia) (General disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (9) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 7 (11) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Rigors, chills (General disorders) | 5 (6) | 0 (0)
Sweating (diaphoresis) (General disorders) | 2 (2) | 0 (0)
Weight loss (General disorders) | 7 (8) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 15 (23) | 2 (2)
Anorexia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 3 (3) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 2 (4) | 0 (0)
Febrile neutropenia (Infections and infestations) | 17 (19) | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 12 (14) | 3 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Glucose, serum-low (hyperglycemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 12 (14) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Mental status (Nervous system disorders) | 1 (1) | 0 (0)
Mood alteration (Nervous system disorders) | 2 (3) | 0 (0)
Neuropathy: cranial (Nervous system disorders) | 1 (1) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 4 (4) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Eyelid dysfunction (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 13 (15) | 0 (0)
Vision-blurred vision (Eye disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 17 (60) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Urinary retention (including neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 16 (19) | 3 (4)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No